CLINICAL TRIAL: NCT04857229
Title: Do the Results of Intra-operative Margin Assessment Correlate With the Output of Conventional Histology for Patient Undergoing Breast Conservation Surgery?
Brief Title: Histolog Comparison to Standard Histology
Acronym: HiCoSH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: SamanTree Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 20CX6399
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Margins of Excision; Breast Cancer
MeSH Terms: conditions — Margins of Excision; Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patient: All recruited patient will have their margins assessed with the confocal microscope with comparison of accuracy against gold standard histology.
  Interventions: Device: Histolog Scanner

INTERVENTIONS:
Device: Histolog Scanner — Confocal Microscope

SUMMARY:
This is a clinical device trial to assess the accuracy of margin assessment for a confocal scanning device (Histolog Scanner) at assessing the margins of breast tissue following wide local excision surgery.

DETAILED DESCRIPTION:
Currently a 15-20% of breast cancer patients have cancer cells seen at the edge of the tissue removed following. These patient will need to undergo a second operation to ensure all the cancer cells are removed, which has psychological, cosmetic and cost implications. Several technologies have been designed to allow the edges of tissue to be tested during surgery, with the most accurate being those that involve assessing the tissue edge at a cellular level. However, these techniques are time consuming which makes their use in routine work impractical.

The Histolog system uses pinhole (confocal) microscopy to capture cellular level images of the edge of tissue intra-operatively. The first generation of the device has been shown to be accurate for assessing breast tissue biopsies and skin cancer. The second generation of the device has an 8cm plate for scanning tissue and is CE marked for the assessment of tissue margins. This project is to show that the device is accurate for the assessment of margins, with further assessment in relation to the time for images to be captured and ease of interpretation to assess overall feasibility. The study would recruit at a single high volume breast cancer centre. The study will recruit patients with a diagnosis of breast cancer who are due to undergo breast conservation surgery (lumpectomy) with inclusion criteria of female patients over the age of 18 who are able to give informed consent. The study would involve the edges of removed tissue being imaged following surgery. These images would be reported by a consultant histopathologist and compared to the routine gold standard histology. There is no change to patient care and the device will not be used to change the surgery performed. There are no questionnaires or additional demands placed on the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of providing informed consent
* Female
* Have a diagnosis of invasive breast cancer or ductal carcinoma in-situ
* Have been discussed within the multidisciplinary meeting with a recommendation that the patient is suitable for breast conservation therapy
* Any localisation technique can be used of impalpable lesions (eg if the wire impairs the image quality, this will inform for full scale research)
* Patient undergoing breast conservation surgery
* Patient undergoing further breast conservation surgery for positive margins after previous surgery
* Patient's will be able to participate for a re-excision of margin, even if they did not participate for their initial operation

Exclusion Criteria:

Patient undergoing mastectomy, including completion mastectomy due to involved margins

* Patients undergoing excision biopsies
* Male patients
* Patients under the age of 18
* Unable to provide valid consent in English language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing surgery for breast cancer, who are due to undergo breast conservation surgery. Patient with a diagnosis of invasive breast cancer or DCIS are eligible for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To compare the sensitivity and specificity of involved margins being assessed intra-operatively using Histolog® Scanner system against conventional histology reporting for patient undergoing breast conservation surgery for breast cancer. | 6 months
  To compare the sensitivity and specificity of involved margins being assessed intra-operatively using Histolog® Scanner system against conventional histology reporting for patient undergoing breast conservation surgery for breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Leff, MBBS FRCS (Gen Surg) MS PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No